CLINICAL TRIAL: NCT05323539
Title: Comparison of Thyroid Volumes by Ultrasonography in Patients With and Without Endometrioma
Brief Title: Comparison of Thyroid Volumes in Patients With and Without Endometrioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulsum Uysal, Associate Professor Gulsum Uysal, Adana City Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1557/2021
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Endometrioma; Thyroid
MeSH Terms: conditions — Endometriosis; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with endometrioma (Active Comparator): Patients having a prediagnosis of surgically planned endometrioma occured this group.
  Interventions: Other: Evaluating Thyroid Volumes by ultrasonography
- Control group (Active Comparator): Patients who had planned gynecological surgery for a reason (ovarian cycts) other than endometrioma
  Interventions: Other: Evaluating Thyroid Volumes by ultrasonography

INTERVENTIONS:
Other: Evaluating Thyroid Volumes by ultrasonography — The inclusion criteria are ; having a prediagnosis of surgically planned endometrioma and to undergo gynecological surgery for a reason other than endometriosis (control group). Among the patients with pre-diagnosis of endometriosis, who applied to our clinic during the study period and accepted to participate in the study, thyroid volumes will be measured by ultrasonography during the preoperative hospitalization. The pathological diagnosis of the patients will be confirmed and patients with different results will be excluded from the study (such as malignancy, endometriosis prediagnosis but different pathology detected etc.) In the same period, gynecological surgery was planned for another reason and patients without endometriosis will form the control group.
  Other Names: routine blood tests, pathology data reports

SUMMARY:
The aim of our study is to evaluate whether there is a statistical difference between thyroid gland volume in patients with pathological diagnosis of endometriosis or endometrioma and in patients who underwent surgery for other gynecological reasons, and to reveal the presence of concomitant thyroid disease in these cases.

DETAILED DESCRIPTION:
Transcripts and proteins involved in thyroid metabolism are dysregulated in the eutopic and ectopic endometrium of endometriotic patients, leading to triiodothyronine (T3) action, resistance, and local thyroxine (T4) accumulation of the ectopic endometrium. Thyroid stimulating hormone (TSH) acts as a proliferative and prooxidative hormone in all endometriums of endometriosis patients and controls. Mouse studies have confirmed that endometriotic implants are larger when thyroid hormones are increased.

Since endometriosis is characterized by a chronic inflammatory process, the high prevalence of autoimmune thyroid diseases in patients with endometriosis may be the result of immune dysregulation observed in women with endometriosis (5). Thyroid involvement has already been described in the physiology of the endometrium and ovary, and thyroid diseases are often associated with gynecological and obstetric disorders such as infertility, miscarriage or preterm delivery.

Despite all the links between thyroid diseases and endometriosis, there is no study related to thyroid volume in patients with endometriosis so far. Thyroid volume was studied in patients with diabetes mellitus, pregnant women, and scleroderma. We believe that the evaluation of thyroid volume in patients with endometriosis will contribute to the investigation of the relationship between these two pathogenesis, and to the treatment and follow-up approach.

ELIGIBILITY:
Inclusion Criteria:

* Prediagnosis of surgically planned endometrioma

Exclusion Criteria:

* Patients with goiteri,
* Patients with past or present autoimmune thyroid dysfunction,
* Patietns on treatment with thyroid hormones or drugs containing iodine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — having a prediagnosis of surgically planned endometrioma
Enrollment: 60 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Measuring Thyroid Volumes by ultrasonography | 6 months
  Longitudinal and transverse scans are performed allowing the measurement of the depth, the width and the length of each lobe. The ellipsoid formula is used. The thyroid volume is the sum of the both lobes excluding isthmus. All measurements are performed bt one experienced radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Uysal, Principal Investigator — University of Heath and Sciences Adana City Training and Research Hospital
Locations (1):
- Adana City Education and Research Hospital, Adana, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No